CLINICAL TRIAL: NCT03504085
Title: Mind/Body Interventions for Chronic Low Back and Neck Pain in Military Personnel
Brief Title: Overcoming Pain Through Yoga in the Military
Acronym: OPTYM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Erik Groessl, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34AT009073-01 (NIH); R34AT009073-01 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-04-20 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain
Keywords: Chronic Low Back Pain; CLBP; Chronic Neck Pain; CNP; Chronic Pain; Military; Active Duty; Yoga; Mindbody
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: We will be conducting a pilot RCT with two types of yoga interventions. A total of 50 participants will be randomized to attend either active Hatha yoga or restorative yoga. Enrollment will be conducted on a rolling basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga (Experimental): This arm will receive the active Hatha yoga intervention. Instructors lead participants through various yoga poses for 60-minutes, 1-2x weekly for 12 weeks, and daily home practice is recommended.
  Interventions: Other: Yoga: Active Hatha
- Restorative Yoga (Active Comparator): This arm will receive a restorative yoga intervention. Instructors guide participants through relaxation exercises, typically with eyes closed, laying down, and minimal movement 60-minutes, 1-2x weekly for 12 weeks.
  Interventions: Other: Yoga: Restorative

INTERVENTIONS:
Other: Yoga: Active Hatha — Classical Hatha yoga with influences from Viniyoga and Iyengar yoga. Both Viniyoga and Iyengar yoga styles emphasize modifications and adaptations including the use of props such as straps and blocks in order to minimize the risk of injury and make the poses accessible to people with health problems and limitations
  Other Names: Active
  Arms: Hatha Yoga
Other: Yoga: Restorative — Restorative Yoga is a slow-paced yoga style that emphasizes relaxation and includes very little movement.
  Other Names: Non-Active
  Arms: Restorative Yoga

SUMMARY:
Our primary aim is to assess the feasibility of conducting yoga research among active-duty military personnel with Chronic Low Back Pain (CLBP) and/or Chronic Neck Pain (CNP). In addition, we will evaluate the yoga intervention preferences and refine an existing yoga intervention to address those needs. The study will prepare us for a R01 funded pragmatic clinical trial of yoga for CLBP and CNP in active-duty military.

DETAILED DESCRIPTION:
In preparation for a full-scale study via a subsequent R01 proposal, our study objective is to examine the feasibility and acceptability of conducting a yoga RCT among active-duty military personnel with CLBP/CNP in military and community settings. The study will be conducted in two phases: Phase 1 (completed) involved obtaining IRB approval to conduct research in military settings, collecting qualitative data from stakeholders on attitudes and preferences for yoga interventions, and refining the existing Yoga for CLBP intervention for the needs of active-duty military and persons with CNP. Phase 2 will recruit and randomize 50 military personnel with CLBP or CNP to either active hatha or restorative yoga. Pain interference, pain severity, physical function, opioid medication use, and mental health outcomes are of primary interest. Mechanisms will also be studied.

The specific aims are as follows:

Aim 1: Evaluate and navigate barriers and facilitators for obtaining IRB approval to conduct randomized controlled intervention studies with active-duty military personnel.

Aim 2: Evaluate the acceptability of and preferences for yoga interventions among active-duty military personnel with CLBP/CNP.

Aim 3: Refine and modify the existing Yoga for CLBP intervention to address CNP, and the needs of active-duty military personnel.

Aim 4: Evaluate the feasibility of recruitment of active-duty military personnel with CLBP/CNP into a yoga RCT.

Aim 5: Evaluate the adherence of this population to the two yoga interventions. Aim 6: Obtain effect size estimates to inform power analyses for a full-scale RCT.

Accomplishing these aims will prepare us for an R01 proposal to study the efficacy of yoga for military personnel with CLBP/CNP in a full-scale randomized, controlled trial. To be successful and maximize the scientific knowledge obtained from an R01 study, it is crucial to first establish working relationships with military researchers, ensure that recruitment and randomized assignment are feasible, pilot test measurement strategies, and ensure that both interventions will be well-attended and have been optimally chosen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLBP or CNP > 6 months
* Willing to attend a yoga program for 12 weeks
* Willing to complete 3 assessments
* English literacy
* Have had no changes in pain treatments in the past month
* Willing to not change pain treatments during study unless medically necessary
* Have not practiced yoga more than 2x in the last 12 months

Exclusion Criteria:

* Back or neck surgery within the last year
* Back or neck pain due to specific systemic problem (e.g., lupus, scoliosis)
* Severe vertebral disk problems,
* Persistent sciatica or nerve compression > 3 months
* Coexisting chronic pain problem (e.g., migraine headaches, fibromyalgia)
* Serious or unstable psychiatric illness (e.g., psychosis, mania, episode, or substance dependence)
* Major coexisting medical illness (e.g., cancer, COPD, morbid obesity)
* Positive Romberg test (with or without sensory neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Groessl, Ph.D., Principal Investigator — University of California, San Diego; Ian Fowler, MD, Principal Investigator — Navy Medical Center San Diego
Locations (2):
- United States (2):
  - UCSD's Health Services Research Center, San Diego, California
  - Navy Medical Center San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groessl EJ, Casteel D, McKinnon S, McCarthy A, Schmalzl L, Chang DG, Fowler IM, Park CL. Comparing Types of Yoga for Chronic Low Back and Neck Pain in Military Personnel: A Feasibility Randomized Controlled Trial. Glob Adv Health Med. 2022 Jun 16;11:2164957X221094596. doi: 10.1177/2164957X221094596. eCollection 2022. PMID 35734420

RESULTS

PARTICIPANT FLOW:
Period: End of Intervention - 12 Weeks
Arm/Group | Hatha Yoga | Restorative Yoga
Started | 24 | 25
Completed | 21 | 21
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4
Period: Final Assessment - 6 Months
Arm/Group | Hatha Yoga | Restorative Yoga
Started | 24 | 25
Completed | 19 | 20
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hatha Yoga | Restorative Yoga | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9.1) | 32 (8.1) | 33 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 21 | 17 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference
Description: Brief Pain Inventory (BPI) : Self-Report measure of pain interference and pain severity consisting of 14 items. The measure includes front and back body diagrams to describe areas of pain, four pain severity items and seven pain interference items rated on 0-10 scales, and one question about percentage of pain relief by analgesics. The pain interference score is the mean of the 7 interference items. The pain severity score is the mean of 4 severity items.
  Scale scores are the mean of relevant items. Thus, scores range from 0-10 with higher scores indicating more pain interference.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: Effect size
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 4.2 (2.2) | 4.0 (2.4)
  12 weeks | 3.9 (2.4) | 3.2 (2.5)

2. Secondary Outcome: Roland-Morris Disability Questionnaire
Description: Self-report measure consisting of 23 questions that ask about limitations experienced for a variety of daily activities.
  Scale scores are the sum of items endorsed, thus scores range from 0-23 with higher scores indicating more back pain-related disability.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 10.8 (5.2) | 10.0 (5.6)
  12 weeks | 10.1 (6.3) | 7.6 (6.1)

3. Secondary Outcome: BPI Pain Severity
Description: Brief Pain Inventory (BPI) : Self-Report measure of pain severity consisting of 4 items. The measure includes front and back body diagrams to describe areas of pain, four pain severity items and seven pain interference items rated on 0-10 scales, and one question about percentage of pain relief by analgesics. The pain severity score is the mean of 4 severity items.
  Scale scores are the mean of relevant items. Thus, scores range from 0-10 with higher scores indicating greater pain severity.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes - Cohen's d
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 4.7 (1.7) | 4.7 (1.8)
  12 weeks | 4.0 (2.3) | 3.7 (1.9)

4. Secondary Outcome: Neck Disability Index
Description: Ten-item self-report measure to assess neck pain interference in daily life activities.
  Each of the 10 items is scored from 0 - 5. The items are summed and scores range from 0-50 with higher scores indicating greater disability due to neck pain.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 14.3 (9.3) | 12.1 (9.0)
  12 weeks | 14.0 (10.7) | 10.0 (8.9)

5. Other Pre Specified Outcome: Health Related Quality of Life (HRQOL) Short-form 12 (SF12) - Physical
Description: 12-Item self-report measure on individual's views about their physical health.
  Scores are scaled to range from 0-100 with higher scores indicating better physical quality of life.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 33.1 (7.3) | 36.5 (10.5)
  12 weeks | 37.0 (8.1) | 39.2 (9.6)

6. Other Pre Specified Outcome: HRQOL - SF12 - Mental Health
Description: Mental Component Score for the SF12
  Scores are scaled to range from 0-100 with higher scores indicating better mental quality of life.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 47.1 (11.6) | 49.5 (9.5)
  12 weeks | 45.2 (12.5) | 47.1 (10.6)

7. Other Pre Specified Outcome: The Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Scale (FSS) assesses the impact and severity of fatigue with 9 items. A score of > 4.0 constitutes severe fatigue.The measure has good psychometrics for pain disorders.
  This is a 9-item questionnaire with questions related to how fatigue interferes with certain activities and severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score indicate greater fatigue severity.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 4.0 (1.4) | 4.0 (1.5)
  12 weeks | 4.4 (1.6) | 3.8 (1.6)

8. Other Pre Specified Outcome: CES-D 10
Description: Ten-item self-report measure on the frequency of mood symptoms. Scores greater than or equal to 10 indicate depression.
  The 10 items are rated on a Likert scale from 0-3. Thus the total score ranges from 0-30 with higher scores indicating more depression.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Reporting Status: Not Posted

9. Other Pre Specified Outcome: AUDIT-C
Description: The AUDIT-C is a 3-item alcohol screen that reliably identifies patients who are hazardous drinkers or have alcohol use disorders. The AUDIT-C is a modified version of the 10 question AUDIT instrument.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Dimensions of Anger Reactions (DAR)
Description: Developed by Forbes et al., The Dimensions of Anger Reactions questionnaire consists of 7 items and has demonstrated strong internal reliability and concurrent validity with other existing measures of anger.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: The Brief Resilience Scale (BRS)
Description: The Brief Resilience Scale (BRS) assesses and individuals ability to recover from stress or trauma. The measure consists of six items and has good reliability and validity.
  The score is the mean of the 6 items, which are rated from 1 to 5. Scores range from 1-5.0 and higher scores indicate greater resilience.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Self Efficacy for Chronic Low Back Pain Scale
Description: A 6-item self-report measure of an individual's confidence in performing certain activities. Items range from 1 (not at all confident) to 10 (totally confident).
  The score is the mean of the items and ranges from 1-10 with higher scores indicating greater self-efficacy.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Physical Measures: Grip Strength
Description: Grip strength will be measured with a hydraulic dynamometer. Two trials will be performed for each hand and the best performance will be taken for each side. The average of both hands is used for analysis.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Physical Measures: Core Stabilization
Description: Prone and supine bridge positions will assess core stabilization. Participants begin on their elbows in the prone position with shoulders, hips, and ankles aligned. The supine position is tested next, with knees flexed 90 degrees and pelvis raised from the floor with shoulders, hips, and knees aligned. Assessors record length of time (120 seconds max) that each position is held in proper form.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Physical Measures: Balance
Description: Balance will be measures performance on a one-leg stand on each side. Assessors record length of time (2 minutes max) that each one-leg stand is held in proper form.
Time Frame: baseline, 12-weeks, 6-months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: PROMIS - Pain Intensity
Description: PROMIS (Patient-Reported Outcomes Measurement Information System) measure - Pain Intensity
  The PROMIS Pain Intensity instrument consists of three items with 5 response options ranging from 1 ("had no pain") to 5 ("very severe") addressing how much pain the person experiences now and in the past 7 days. The raw score is the sum of the three questions, with a minimum of 3 and a maximum score of 15, with higher scores indicating greater pain intensity.
Time Frame: assessed at baseline, 12 weeks, and 6 months; baseline and 12 weeks reported
Population: effect sizes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Restorative Yoga
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 9.8 (1.7) | 9.5 (2.3)
  12 weeks | 9.0 (2.4) | 8.6 (2.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Hatha Yoga | Restorative Yoga
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 2/24 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=24) | Restorative Yoga (N=25)
leg surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant had an surgey on their leg and could not attend yoga. Event was unrelated to the intervention.
Broken foot or ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Unrelated to yoga intervention.
Back surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Surgery unrelated to intervention
Unspecified surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Injured their shoulder during military training activity. Unrelated to yoga.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03504085/Prot_SAP_000.pdf